CLINICAL TRIAL: NCT04548804
Title: Better Mechanistic Understanding of and Risk Stratification for Ventricular Tachyarrhythmias Through ECGI
Acronym: BREACH-ECGI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: METC19-065; NL69831.068.19 (Other: Toetsingonline); 300260 (Other: Raad van Bestuur)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Ventricular Tachycardia; Ventricular Arrythmia; Ventricular Fibrillation; Polymorphic Ventricular Tachycardia; Sudden Cardiac Death; Sudden Cardiac Arrest; Sudden Cardiac Death Due to Cardiac Arrhythmia; Heart Arrest; Cardiac Death; Cardiac Arrest; Cardiac Arrhythmia; Congenital Heart Disease
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Arrest; Death; Arrhythmias, Cardiac; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Both groups (control and diseased) will undergo a body surface potential mapping and a cardiac + low dose CT-scan.
Who Masked: Care Provider
Masking Description: The treating physician is not informed about the results of the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Control subjects receiving body-surface potential mapping (BSPM) and either a CT-scan or a CMR scan
  Interventions: Diagnostic Test: ECG-Imaging
- Diseased (Experimental): Diseased subjects receiving body-surface potential mapping (BSPM) and either a CT-scan or a CMR scan. Outcome measures from these procedures will be compared to controls.
  Interventions: Diagnostic Test: ECG-Imaging

INTERVENTIONS:
Diagnostic Test: ECG-Imaging — A body surface potential mapping and a cardiac + low dose CT-scan

SUMMARY:
This study aims to evaluate the electrophysiological properties of the heart conduction system in patients with (increased risk of) ventricular tachyarrhythmias (VTA) and sudden cardiac arrest, and in a control cohort. The electrophysiological properties will be measured with the relatively new technique ECG-Imaging (ECGI). Moreover, clinical data of subjects will be gathered.

By combining the data from the data gathering and the results of ECGI, the investigators hope to increase mechanistic understanding of and risk stratification for VTAs. The investigators aim to be able to identify patients at risk of an arrhythmic event, and aim for better treatment strategies in the future.

DETAILED DESCRIPTION:
ECGI combines electrical body-surface mapping with 256 electrodes placed on the thorax with a CT-scan obtaining the anatomy of the heart and torso, hereby able to reconstruct local electrograms, activation and recovery times. In recent research, ECGI provided numerous extra insights into normal cardiac electrophysiology, but also electrophysiological disorders and disease. The results strongly suggest that ECGI can play a pivotal role in further characterizing arrhythmia mechanisms, therefore could do so for VTAs, leading to diagnosis and treatment improvement. Moreover, ECGI seems to have the potential to detect arrhythmogenic substrate in individuals before their first event, offering the possibility to diagnose and treat patients before sudden cardiac arrest occurs.

In the BREACH-ECGI study:

ECGI will be used to noninvasively characterize the epicardial electrophysiological substrate and triggers of:

* Patients with (increased risk of) VTAs
* A control cohort. Results will be evaluated for increased mechanistic understanding and risk stratification.

Moreover, clinical data of subjects will be gathered. These data will be analyzed to determine their prognostic value in terms of arrhythmia risk

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be ≥ 18 years old, have either a history of VTAs or be at risk of VTAs and have one of the following diagnoses:

* Ischemic cardiomyopathy
* Non-ischemic cardiomyopathy
* Non-structural heart disease
* Congenital heart disease (with a limitation to CCTGA and situs inversus)

Or: a subject must be ≥ 18 years old and have a structurally normal heart with a clinical indication for a cardiac CT.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* A known strong reaction against electrode attachment or contrast agent.
* Any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study.
* Pregnancy, nursing or planning to be pregnant.
* The subject has an estimated glomerular filtration rate (eGFR) of <30mL/min/1.73m2, using the MDRD calculation 14.
* Being unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
ECG-Imaging outcome: epicardial potentials | 3 years
  reconstructed epicardial potentials, represented in mV over time(s).
ECG-Imaging outcome: activation and repolarization maps | 3 years
  Activation and repolarization maps. Acivation and repolarization times are determined from the epicardial potentials, expressed in ms. These are shown on a CT-derived or CMR-derived heart mesh. The entire activation and repolarization of the epicardium of the heart can be visualized this way.

SECONDARY OUTCOMES:
(Possible) Prognostic risk factors for recurrent ventricular arrhythmias | 6 years
  Possible risk factors, found in the clinical data collection, expressed as odds/hazard ratio.
Recurrence of ventricular arrhythmias | 6 years
  Documentation over the period of follow-up, if subjects had a recurrence of ventricular arrythmia(s), presented as number of events over a time period.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Jessa Hospital, Hasselt, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: Undecided